CLINICAL TRIAL: NCT03251014
Title: The Thrombotic Effects of Yellowstripe Scad (YSS) Compared to Salmon Among Healthy Overweight Subjects: A Randomized Cross Over Trial
Brief Title: Thrombotic Effects of Yellowstripe Scad
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Collaborators: Ministry of Science, Technology and Innovation (MOSTI) Malaysia (Unknown)
Responsible Party: Principal Investigator, Dr. Loh Su Peng, Associate Professor, Universiti Putra Malaysia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 06-01-04-SF2310; NMRR-16-2693-32300. (Registry Identifier: National Medical Research Register); FPSK(FR16)P005 (Other: Universiti Putra Malaysia)
Record Dates: First submitted 2017-05-30; First posted 2017-08-16 (Actual); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Thrombosis
Keywords: Thrombosis; Yellowstripe scad; Salmon; Healthy overweight subjects; Randomized crossover trial
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YSS/salmon group (Experimental): YSS followed by salmon
  Interventions: Other: YSS; Other: Salmon
- Salmon/YSS group (Experimental): Salmon followed by YSS
  Interventions: Other: YSS; Other: Salmon

INTERVENTIONS:
Other: YSS — Intervention providing steamed whole YSS (~265 g/day, 3 days/week) for eight weeks
Other: Salmon — Intervention providing steamed salmon fillet (~246 g/day, 3 days/week) for eight weeks

SUMMARY:
The study aimed to determine the thrombotic effects of YSS compared with salmon among healthy overweight subjects. It hypothesized that YSS may result significant, favorable thrombotic effects and the effects may be similar with salmon.

DETAILED DESCRIPTION:
The project was a randomized, two-period, crossover trial with 8-week treatment periods and 8-week washout period. A total of 50 healthy overweight adults were recruited among staff and students in UPM. All the subjects were randomized into two groups. Each group was served with either cooked YSS (~265 g/ day) or salmon (~246 g/day) thrice per week. Blood and urine samples were collected for laboratory assessment.

ELIGIBILITY:
Inclusion Criteria:

* Malaysian
* Overweight participants (BMI 23-27.4 kg/m2)

Exclusion Criteria:

* Regular use of fish oil supplements during the last one month
* Regular consumption of fish twice or more per week
* Vegetarian who excluded all meat, fish, and poultry from their diet
* Diagnosed with cardiovascular disease, haemostasis disorder, inflammatory disease, diabetes mellitus, hypertension, or other significant medical history that may prohibits the participation
* Receiving warfarin or aspirin treatment, or medication to lower serum lipids, blood pressure, and inflammation
* Women who are menopause, pregnant or lactating

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-05-09 (Actual); Study Completion 2017-05-09 (Actual)

PRIMARY OUTCOMES:
Changes in hemostatic status assessed by immunoassay method | 8 weeks
  Hemostatic markers including vWF-A2 and CD62b (p-selectin) in pg/mL are evaluated.

SECONDARY OUTCOMES:
Changes in lipid and glucose profiles analysed by medical diagnostic laboratory | 8 weeks
  Total cholesterol, triglyceride, HDL-cholesterol, LDL-cholesterol, VLDL-cholesterol, and fasting blood glucose in mmol/L are evaluated.
Changes in liver enzymes analysed by medical diagnostic laboratory | 8 weeks
  Serum levels of alanine transaminase (ALT), aspartate transaminase (AST), alkaline Phosphatase (ALP) and gamma glutamyl transferase (GGT) in IU/L are determined.
Changes in renal function analysed by medical diagnostic laboratory | 8 weeks
  Serum levels of creatinine, urea, and electrolytes (sodium, potassium, and chloride) in mmol/L are determined.
Changes in body mass index (BMI) | 8 weeks
  Weight and height are combined to report BMI in kg/m^2
Changes in blood pressure | 8 weeks
  Seated systolic and diastolic blood pressures are taken in mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Su Peng Loh, PhD, Principal Investigator — Universiti Putra Malaysia

IPD SHARING:
Plan to Share IPD: No